CLINICAL TRIAL: NCT00022113
Title: A Phase I Study of EMD 121974 in Patients With Advanced Solid Tumors
Brief Title: EMD 121974 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02392; 00-1096; U01CA099176 (NIH); CDR0000068786 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Cilengitide

ARMS (1):
- Treatment (cilengitide) (Experimental): Patients receive EMD 121974 IV over 1 hour twice weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cilengitide; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cilengitide — Given IV
  Other Names: EMD 121974
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of EMD 121974 in treating patients who have advanced solid tumors. EMD 121974 may slow the growth of solid tumors by stopping blood flow to the tumor

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the toxic effects and maximum tolerated dose of EMD 121974 in patients with advanced solid tumors.

II. Determine the biologic activity of this drug in these patients. III. Determine the pharmacokinetic profile and plasma biological effects of this drug and identify any relationship with its biologic activity or observed toxicity in these patients.

IV. Determine, preliminarily, the antitumor efficacy of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive EMD 121974 IV over 1 hour twice weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-10 patients receive escalating doses of EMD 121974 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor that is refractory to standard therapy or for which no standard therapy exists
* Tumors must be amenable to minimally-invasive biopsy (i.e., tumors must be superficial enough to be sampled by punch biopsy or core biopsy procedure without radiologic guidance)*
* No uncontrolled brain metastases, including symptomatic lesions or lesions requiring glucocorticoids and/or anticonvulsants to suppress symptoms

  * Negative brain scan required if there are signs and symptoms suggestive of brain metastasis
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* At least 12 weeks
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL
* Bilirubin normal
* AST and ALT no greater than 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No ongoing or active infection
* No other concurrent serious systemic disorders (e.g., significant CNS illness) that would preclude study
* No concurrent psychiatric illness or social situations that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent anticancer immunotherapy
* Concurrent hematologic growth factors for cytopenias allowed
* At least 4 weeks since prior anticancer chemotherapy (6 weeks for nitrosoureas, carmustine, or mitomycin) and recovered
* See Disease Characteristics
* No concurrent anticancer hormonal therapy
* Concurrent oral contraceptives or postmenopausal hormone replacement allowed
* Recovered from prior radiotherapy
* At least 2 weeks since prior palliative radiotherapy to bone or brain metastases
* At least 4 weeks since prior anticancer radiotherapy
* No concurrent anticancer radiotherapy
* Not specified
* At least 4 weeks since prior anticancer therapy and recovered
* At least 4 weeks since prior investigational agents
* Any number of prior therapies allowed
* No other concurrent anticancer investigational or commercial agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2001-05; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
MTD of cilengitide defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. | 4 weeks
  Graded according to the NCI Common Toxicity Criteria version 2.0.
Toxic effects of cilengitide described as an adverse event that has an attribution of possibly, probably or definitely related to investigational treatment | Up to 4 years
  Graded according to the NCI Common Toxicity Criteria version 2.0.
Biological activity of this regimen | Up to 4 years
  Measured buy TUNEL assay, CD31 immunohistochemistry, dynamic contrast-enhanced MRI, and FDG-PET scan.

SECONDARY OUTCOMES:
Pharmacokinetics of cilengitide | At 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 8.0, and 24.0 hours post-end-of-infusion on day 1 of course 1
Observation of response consisting of complete response, partial response, or stable disease, evaluated using the RECIST criteria | Up to 4 years
Time to progression | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Michele Basche, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Colorado, United States